CLINICAL TRIAL: NCT01727986
Title: Extension, Open-label, Interventional, Long-term Study to Evaluate the Safety of Tocilizumab Treatment in Patients From Brazil With Polyarticular-course Juvenile Idiopathic Arthritis Who Completed the Global Multinational Trial (WA19977)
Brief Title: An Extension Long-Term Study of RoActemra/Actemra (Tocilizumab) in Patients With Polyarticular Juvenile Idiopathic Arthritis Who Completed The WA19977 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ML28413
Record Dates: First submitted 2012-11-08; First posted 2012-11-16 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

ARMS (1):
- RoActemra/Actemra (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg or 10 mg/kg iv every 4 weeks, 104 weeks

SUMMARY:
This long-term, open-label extension study will evaluate the safety of RoActemra/Actemra (tocilizumab) in patients with polyarticular-course juvenile idiopathic arthritis who completed the WA19977 core study. Patients aged 9-18 years with at least JIA ACR30 clinical response to RoActemra/Actemra in the core study will be eligible to receive RoActemra/Actemra 8 mg/kg intravenously every 4 weeks. Anticipated time on study treatment is 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients 9 to 18 years of age who completed visit 33 (week 104) of WA19977 study with at least JIA ACR30 clinical response to RoActemra/Actemra relative to baseline in WA19977, with no AEs, SAEs or conditions that lead to unacceptable risk of continued treatment
* Females of child-bearing potential and males with female partners of child-bearing potential must agree to use effective contraception as defined by protocol

Exclusion Criteria:

* Patients with, according to investigator judgment, not satisfactory benefit from RoActemra/Actemra therapy within WA19977
* Treatment with any investigational agent since the last administration of study drug in the core study WA19977 or current participation in another clinical trial except WA19977
* Patient developed any other autoimmune rheumatic disease or overlap syndrome other than the permitted polyarticular-course JIA subsets: rheumatoid factor positive or negative JIA or extended oligoarticular JIA
* Patient is pregnant , lactating, or intending to become pregnant during the study and up to 12 weeks after the last administration of study drug
* Any significant concomitant disease or medical or surgical condition
* History of significant allergic or infusion reactions to prior biologic therapy
* Currently active primary or secondary immunodeficiency
* Current abuse of alcohol, drugs or chemical abuse
* Known and currently active acute, subacute, chronic infections or history of recurrent infection; patients suffering from ongoing active infections with Epstein Barr virus, herpes zoster or recurrent history of urinary tract infection can be included after the (acute) infection has been excluded or subsided
* Positive for latent tuberculosis (TB)
* Currently active asthma for which the patient has required the use of oral or parenteral corticosteroids for >/= 2 weeks within 6 months prior to entering the study
* Inadequate hepatic, renal or bone marrow function

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Long-term safety: Incidence of adverse events | approximately 3 years

SECONDARY OUTCOMES:
Response rates according to the American College of Rheumatology criteria for juvenile idiopathic arthritis (JIA ACR) | approximately 3 years
Proportion of patients achieving inactive disease/clinical remission | approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Brazil (3):
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo